CLINICAL TRIAL: NCT06568549
Title: Reduced Immunosuppression in Older Renal Transplant Recipients With Trugraf® Monitoring (RIOT Trial): A Prospective, Randomized, Multicenter Trial.
Brief Title: Reduced Immunosuppression in Older Renal Transplant Recipients With Trugraf®/TRAC Monitoring (RIOT Trial): A Prospective, Randomized, Multicenter Trial.
Acronym: RIOT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Transplant Genomics, Inc. (Industry); Eurofins (Industry)
Responsible Party: Principal Investigator, Mark Stegall, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-002574
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation; Mycophenolate Mofetil
Keywords: Kidney Transplant
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-Randomized Group (No Intervention): Individuals who do not meet eligibility for randomization will continue in the study and continue to follow study related visits. Individuals will continue with their current immunosuppression medication.
- MMF Maintenance Group (Active Comparator): Individuals randomized to the MMF Maintenance Group will not be withdrawn from their MMF and will continue to follow their standard of care immunosuppression medications.
  Interventions: Drug: Mycophenolate Mofetil (MMF) Maintenance Group
- MMF Withdrawal Group (Experimental): Individuals randomized to the MMF Maintenance Group will be withdrawn from their MMF immunosuppression medication from Month 4 to Month 10 post-transplant.
  Interventions: Drug: Mycophenolate Mofetil (MMF) Withdrawal Group

INTERVENTIONS:
Drug: Mycophenolate Mofetil (MMF) Maintenance Group — Mycophenolate Mofetil (MMF), administered orally as standard of care post kidney transplant as part of their immunosuppression regimen. Maintenance in Immunosuppression medication.
  Other Names: CellCept
  Arms: MMF Maintenance Group
Drug: Mycophenolate Mofetil (MMF) Withdrawal Group — Mycophenolate Mofetil (MMF), administered orally as standard of care post kidney transplant as part of their immunosuppression regimen. Withdrawal of MMF immunosuppression medication.
  Other Names: CellCept
  Arms: MMF Withdrawal Group

SUMMARY:
The purpose of this research is to determine the safety and efficacy of withdrawing MMF (Mycophenolate Mofetil) in kidney transplant recipients who are 55 years or older at the time of receiving a kidney transplant. We are comparing them to patients who receive the standard of care Mycophenolate Mofetil.

DETAILED DESCRIPTION:
Participation will be two years and it involves blood collection, collection of medical information and images from standard of care kidney biopsies. Subjects will be asked to complete questionnaires for the study at 12 and 24 months after kidney transplant. The research blood tests that are being collected for the study are called Trugraf®, Eurofins TRAC®, Trac-ID and Immunophenotyping and Single Cell RNA -sequencing. The principal investigator is using this test to see if they can predict and monitor rejection and viral infections in our kidney transplant patients. Immunophenotyping and single cell RNA sequencing tests are being done to identify unique gene expression profiles and their functions in different immune cells.

At the time of the 4 month standard of care kidney biopsy, if participants have not experienced any rejection episodes or formed any donor specific antibodies (dnDSA) and are still eligible, randomization will occur. Participants will be put into 1 of 2 groups: Mycophenolate Mofetil Maintenance group where the subject would continue on current medication, or the subject will be placed into the MMF Withdrawal group which means they would slowly be withdrawn from this medication. If the subject is not eligible to be randomized, they will remain in the study and placed into the Non-Randomized group and continue to have study related visits and procedures like the MMF Maintenance group.

ELIGIBILITY:
Inclusion Criteria:

* Solitary kidney transplant recipient >55 years of age. At most 1 prior solitary kidney transplant.
* No other solid organ transplant though recipients of autologous stem cell transplants are eligible.
* HIV negative.
* Subjects must be on tacrolimus and mycophenolate mofetil or Myfortic at the time of consent. Prednisone at the time of consent is optional and is per local standard of care. Patients randomized to MMF withdrawal will be placed on prednisone 5mg/d at 4 months. Use of other immunosuppression medications for maintenance (cyclosporine, azathioprine, belatacept, sirolimus) is excluded.

Exclusion Criteria:

Time of Transplant Exclusion Criteria:

* The results of the most recent DSA testing indicate DSA with an MFI >2000.
* The results of the most recent cPRA testing indicate cPRA is above >80% (based on MFI >2000).
* Has a history of an underlying clinically significant acute or chronic medical condition or physical examination findings which, in the opinion of the investigator, would make study participation not in the participants best interest (e.g. compromises their well-being) or that could prevent, or limit the protocol specified assessment.

  4-Month Exclusion Criteria:
* Acute rejection episode either clinical or on biopsy (greater than borderline). Subjects must not experience any type of rejection episodes from the time of transplant and must not show any signs of rejection (Cellular or Antibody mediated rejection, excluding borderline) at their 4-month standard of care biopsy Subjects experiencing rejection will not be eligible for randomization and MMF withdrawal.
* Subjects who are unable to undergo their 4-month standard of care kidney biopsy due to medical contraindications.
* De novo DSA
* Subjects who are not maintained on tacrolimus, mycophenolate mofetil of Myfortic. Subjects who are not on tacrolimus and mycophenolate mofetil or Myfortic at the time of randomization will be placed in the non-randomized group.
* Has a history of an underlying clinically significant acute or chronic medical condition or physical examination findings which, in the opinion of the investigator, would make study participation not in the participants best interest (e.g., compromise the well-being) or that could prevent, or limit the protocol-specified assessment.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute Rejection | 4 to 24 months post transplant.
  Total number of subjects to experience acute rejection of the renal transplant
Patient Deaths | 4 to 24 months post transplant.
  Total number of subject deaths from 4-24 months post transplant.
Graft Failure | 4 to 24 months post transplant.
  Total number of subjects to experience graft failure from the renal transplant

SECONDARY OUTCOMES:
Serious Adverse Events (SAE) | 1 and 2 years post transplant.
  The total number of subjects to experience SAE's. Defined as subjects experience any one of the following: acute cellular or antibody medicated rejection, borderline rejection or dnDSA (De novo donor-specific antibodies)
eGFR (estimated glomerular filtration rate) | 2 years post transplant
  eGFR is calculated from a lab blood test using a formula that measures the level of creatinine. In this test a higher number is better. An eGFR value lower than 60 is a sign that the kidneys may not be working properly. Measured as mL/min/1
Single antigen beads (SAB) for donor-specific antibodies | Baseline, 1 year post transplant and 2 years post transplant
  Single antigen bead (SAB) assay is a lab blood test used to detect human leukocyte antigen antibodies (HLA) and assessing the immunological risk for organ transplant. For HLA-DRβ1/3/4/5 the single molecule mismatches can range from 0-22 and for HLA-DQα1/β1 the single molecule mismatches range from 0-31. Measured as pg/mL.
BANFF scores | 2 years post transplant.
  The Banff 2018 classification involves scoring numerous characteristics of renal biopsy specimens. The scores can take values of 0, 1, 2, or 3 for each characteristic, indicating increasing severity of disease as the scores increase.
Absolute lymphocyte counts | 1 year post transplant and 2 years post transplant
  An absolute lymphocytes count is determined by multiplying the total number of white blood cells by the percentage of white blood cells that are lymphocytes. The normal range for lymphocytes is between 800 and 5000 (0.8-5.0) lymphocytes per mL of blood. A normal lymphocytes percentage is 18-45% of total white blood cells. Measured as cells per microliter (cells/µL)
Transplant Related Symptom (CIRS) Questionnaire | 2 years post transplant.
  The CIRS questionnaire is a 36-item questionnaire that contains statements that rate transplant symptoms on a scale of 1(None) to 5 (Very Severe). Total scores range from 36-180, lower scores indicate less severe symptoms, higher scores indicate more severe symptoms.
Albumin/Creatinine Ratio (Microalbumin) Urine | 2 years post transplant
  The urine albumin-creatinine ratio (uACR) test measures the amount of two different substances in urine - albumin (a protein) and creatinine. A value of 30 or higher suggests a higher risk for kidney failure. Measured as mg/g

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Plans for data sharing may include data summaries consisting of tables, charts, and figures. Data included will be anonymous and could include demographics, clinical data collected during the study and correlations with Trugraf and Viracor results. Aggregate data for demographics, Subject ID, etc. will only be shared for involving of milestones.
  The clinical study final report and paper submitted for any publication will also be submitted.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Ongoing data analysis will be performed throughout the study. After completion of all study subjects' visits, final data will be cleaned, reviewed and analyzed by study staff. A clinical summary report would be expected to be delivered to TGI-Eurofins within a year of subject completed visits. We would expect a paper to be written and submitted to a journal for review and acceptance within 2 years of final study completion.
Access Criteria: Data sharing with TGI- Eurofins and study staff.